CLINICAL TRIAL: NCT00987116
Title: Comparison of Two Tapering Strategies of Prednisone in Patients With Generalised Myasthenia Gravis Treated With Prednisone and Azathioprine: a Single-blind Randomised Controlled Multicenter Study
Brief Title: Study Comparing Two Tapering Strategies of Prednisone in Myasthenia Gravis
Acronym: MYACOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P051055
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia gravis; Steroids side effects; Comparison of strategies for tapering steroids; Generalized MG corresponding to grade III, IV or V of MGFA
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Starting dose Prednisone Azathioprine (Active Comparator): Classical Strategy
  Interventions: Drug: Prednisone - Azathioprine
- Starting dose Prednisone - Azathioprine (Active Comparator): Rapid strategy
  Interventions: Drug: Prednisone - Azathioprine

INTERVENTIONS:
Drug: Prednisone - Azathioprine — Rapid strategy consists of decreasing the prednisone dose if at each monthly consultation the patient fulfils the criteria for improvement or minimal manifestation state, in order to discontinue it before twelve months. The starting dose is 0.75 mg/kg/day.
  Classical strategy consists of decreasing the prednisone dose if at each monthly consultation the patient fulfils the criteria for minimal manifestation state, in order to discontinue it before twelve months. The starting dose is 1.5 mg/kg/2days.

SUMMARY:
Pathology - Generalized myasthenia gravis (MG) is cause of muscle weakness that can have a significant impact on daily life activity but can also be, when respiratory or bulbar muscles are involved, life-threatening.

Rationale - Additionally to thymectomy, which indication of is still debated in absence of thymoma, the long-term treatment of generalized myasthenia gravis includes usually prednisone and azathioprine. However, the most used scheme for prescribing and tapering corticosteroid in MG resulted in a very important cumulative dose of prednisone. Indeed, at twelve month, more than 50 percent of patients are still daily treated with at least 18 mg of prednisone and the proportion of patients who are in remission and no longer taking prednisone is very low (Palace and NEWSOM Davis, Neurology 1998). Prolonged corticosteroid therapy is accompanied with various and major side effects, hypertension, osteoporosis, weight gain, glaucoma. Therefore, tapering, eventually discontinuing, prednisone earlier is a relevant therapeutic goal.

For this reason, the investigators will compare to the standard one, a strategy consisting of a rapid decrease in corticosteroid.

Objective - To assess whether, in patients with generalized MG requiring a long-term treatment with corticosteroids and azathioprine, that the strategy of rapid tapering allows discontinuing more rapidly the prednisone for equivalent efficacy than the classical strategy.

DETAILED DESCRIPTION:
Rapid strategy consists of decreasing the prednisone dose if at each monthly consultation the patient fulfils the criteria for improvement or minimal manifestation state, in order to discontinue it before twelve months. The starting dose is 0.75 mg/kg/day.

Classical strategy consists of decreasing the prednisone dose if at each monthly consultation the patient fulfils the criteria for minimal manifestation state, in order to discontinue it before twelve months. The starting dose is 1.5 mg/kg/2days.

Duration of follow-up is 15 months.

In both arms, Myasthenia Muscular Score (MMS), activities of Daily Living Scale (ADLS), MGFA Clinical Classification and MGFA Post-Intervention Status as well as prednisone and azathioprine side effects will be monthly assessed by a senior neurologist who will be blind for treatment group. A second physician, who is aware of the patient's therapeutic group, will then prescribe prednisone dose and tapering for a month, according to MGFA Post-Intervention Status.

In case of worsening, prednisone dose will be increased. In case of exacerbation, the patients will be hospitalised for eventually IvIg infusion or plasma exchange. In case of a severe side effect, prednisone will be reduced irrespectively of MGFA Post-Intervention Status. In case of side effect, azathioprine will be replaced by mycophenolate mofetil.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the patient, after informing
* Generalized MG of grade III, IV or V - Classification MGFA
* Follow-up on 15 months possible and accepted by patients

Exclusion Criteria:

* Age<18 or >80 years
* Pregnancy
* Myasthenia of grade I or II of MGFA
* Patients already treated with prednisone or azathioprine
* Contraindication for prednisone or azathioprine
* Other associated disease requiring a treatment with prednisone or azathioprine
* Weight >100kg
* Invasive thymoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have reach minimal manifestation state (according to MGFA criteria) and are not treated with prednisone after 12 months of treatment and have not relapsed during the next 3 months. | 15 months

SECONDARY OUTCOMES:
Cumulative dose of prednisone at twelve months | 15 MONTHS
Proportion of patients having reached minimal manifestation state 12 months | 15 MONTHS
Time for reaching the improvement or minimal manifestation state (MGFA criteria) | 15 MONTHS
Frequency of exacerbations within the first 15 months after randomization | 15 MONTHS
Frequency of treatment by IvIg or plasma exchange within the first 15 months after randomization | 15 MONTHS
Frequency and type of complications related to prednisone. | 15 MONTHS
Frequency and type of complications of azathioprine | 15 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Sharshar, MD PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Raymond Poincaré, Garches, France

REFERENCES:
- [Derived] Sharshar T, Porcher R, Demeret S, Tranchant C, Gueguen A, Eymard B, Nadaj-Pakleza A, Spinazzi M, Grimaldi L, Birnbaum S, Friedman D, Clair B; MYACOR Study Group. Comparison of Corticosteroid Tapering Regimens in Myasthenia Gravis: A Randomized Clinical Trial. JAMA Neurol. 2021 Apr 1;78(4):426-433. doi: 10.1001/jamaneurol.2020.5407. PMID 33555314